CLINICAL TRIAL: NCT04191876
Title: Financial Incentives to Improve Medication Adherence: a Pilot Study
Brief Title: Financial Incentives to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-0739-ZHH
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Bipolar Disorder; Depression
Keywords: financial incentives; medication adherence; severe mental illness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depression; Medication Adherence; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): This study has only one arm. All patients enrolled will take part in the experimental arm.
  Interventions: Other: Wellth - Financial Incentives

INTERVENTIONS:
Other: Wellth - Financial Incentives — Patients who are willing to participate will be offered financial incentives for medication adherence through an app (Wellth) over 10 weeks.

SUMMARY:
Medication adherence is a challenge in all of medicine and is associated with multiple negative outcomes. Strategies to better measure and enhance adherence to medication are urgent and necessary to minimize unwanted health outcomes, hospitalizations, poorer quality of life and excessive costs for individuals, insurers and caregivers. Recently, behavioral economics-based approaches have emerged as a promising tool to address this unmet need, but its effectiveness in oral antipsychotic treatment remains to be assessed. For this project, investigators will use an app that offers financial incentives to increase compliance for patients with chronic diseases. Investigators intend to enroll 25 patients in a pilot project to assess feasibility of offering financial incentives to improve medication adherence in severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

1. Psychiatric patients with suspected or confirmed poor oral medication adherence.
2. Age 18-80 years old
3. English speaking, since the app being used is only available in English
4. Owning a Smartphone, since the app requires a Smartphone to work
5. Willing and able to participate.

Exclusion Criteria:

1. Acute anger to self or others as per investigator assessment
2. Unwilling or unable to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence rate | Between baseline and study completion (10 weeks)
  Adherence rate will be measured as pills missed/pills prescribed

CONTACTS AND LOCATIONS:
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guinart D, Sobolev M, Patil B, Walsh M, Kane JM. A Digital Intervention Using Daily Financial Incentives to Increase Medication Adherence in Severe Mental Illness: Single-Arm Longitudinal Pilot Study. JMIR Ment Health. 2022 Oct 12;9(10):e37184. doi: 10.2196/37184. PMID 36222818